CLINICAL TRIAL: NCT04286243
Title: UNCPM 21904 - Prevention of Cervical Cancer Through an HPV-based Screen-and-treat Strategy in Malawi: a Cluster Randomized Trial
Brief Title: Prevention of Cervical Cancer Through an HPV-based Screen-and-treat Strategy in Malawi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-0638; UNCPM 21904 (Other: University of North Carolina at Chapel Hill)
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2022-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Model 1 involves: 1) cervico-vaginal self-sampling for high-risk HPV (hr-HPV) while waiting for appointments at the VFP clinic or other clinics, 2) same-day VIA for those women found to be hr-HPV-positive by rapid GeneXpert HPV testing, and 3) same-day thermocoagulation treatment for HPV-positive women who are eligible for ablative therapy by VIA.
  Model 2 will offer women the same services as in Model 1, but they will also be given the option to perform cervico-vaginal self-sampling in the community, via Heath Surveillance Assistants (HSAs) who will bring their HPV sample to the clinic and notify them to return to the clinic for VIA and possible same-day thermocoagulation if their hr-HPV test is positive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Model 1 - Clinic Based Screening (Active Comparator): Model 1 involves: 1) cervico-vaginal self-sampling for high-risk HPV (hr-HPV) while waiting for appointments at the VFP clinic or other clinics, 2) same-day VIA for those women found to be hr-HPV-positive by rapid GeneXpert HPV testing, and 3) same-day thermocoagulation treatment for HPV-positive women who are eligible for ablative therapy by VIA
  Interventions: Other: Clinic-based HPV screening strategy
- Model 2 - Community Based Screening (Experimental): Model 2 will offer women the same services as in Model 1, but they will also be given the option to perform cervico-vaginal self-sampling in the community, via Heath Surveillance Assistants (HSAs) who will bring their HPV sample to the clinic and notify them to return to the clinic for VIA and possible same-day thermocoagulation if their hr-HPV test is positive
  Interventions: Other: Community-based HPV screening strategy

INTERVENTIONS:
Other: Community-based HPV screening strategy — Offering HPV self-collection for cervical cancer screening in the community
  Arms: Model 2 - Community Based Screening
Other: Clinic-based HPV screening strategy — Offering HPV self-collection for cervical cancer screening in the clinic
  Arms: Model 1 - Clinic Based Screening

SUMMARY:
The purpose of the study is to determine the acceptability, appropriateness, and feasibility of implementing new strategies to screen and treat eligible women for cervical cancer through a cluster randomized trial of two different models. Both models offer the same screening and treatment algorithm, but one will be based in Voluntary Family Planning (VFP) or other clinics and the second will be based in the community. Participants will be recruited from two districts in Malawi with the highest HIV prevalence in the country: Lilongwe in the Central Region and Zomba in the Southern Region.

DETAILED DESCRIPTION:
Cervical cancer is largely preventable through screening and preventive therapy. This is a cluster randomized trial that will integrate a novel cervical cancer screen-and-treat algorithm into voluntary family planning (VFP) services via two different models aimed at reducing barriers to screening and treatment in resource limited settings. Model 1 involves: 1) cervico-vaginal self-sampling for high-risk HPV (hr-HPV) while waiting for appointments at the VFP clinic or other clinics, 2) same-day visual inspection with acetic acid (VIA) for those women found to be hr-HPV-positive by rapid GeneXpert HPV testing, and 3) same-day thermocoagulation treatment for HPV-positive women who are eligible for ablative therapy by VIA. Model 2 will offer women the same services as in Model 1, but they will also be given the option to perform cervico-vaginal self-sampling in the community via Heath Surveillance Assistants (HSAs) who will bring their HPV sample to the clinic and notify them to return to the clinic for VIA and possible same-day thermocoagulation if their hr-HPV test is positive. Participants will be recruited from 16 high HIV-prevalence clinics in either Lilongwe in the Central Region or Zomba in the Southern Region. The broad objective of the project is to compare the effectiveness and budget impact of these two models for averting potential cervical cancer cases and to evaluate the implementation and acceptability of the models in multiple different health care facility settings.

A systematic Implementation Evaluation will be conducted throughout implementation of the assigned models at the study health facilities to determine the success/failure in the delivery of intervention packages. The study team will employ the following mixed method data collection assessments:

* In-Depth Interviews with purposively selected healthcare facility staff and clients in the sampled facilities (N = approximately 60).
* Focus group discussions (FGDs) with purposively selected in-clinic services providers and HSAs (N = approximately 160).
* Structured weekly observations of service delivery by clinical mentors using an observation checklist, to observe providers and laboratorians adherence to standards, guidelines and intervention protocols.
* Aggregate collection of routine quantitative service utilization data from adapted family planning and cervical cancer screening registers.
* Implementation of assessment tools to assess changes in service providers' workload.
* Client Exit Surveys with women in the catchment areas of the targeted facilities who received or declined family planning and/or cervical cancer screening services at the facility or in the community (N= approximately 1,000).
* Time and motion studies to observe visits and staff time spent on counseling, screening and treatment procedures, and managing and testing specimens.

Finally, an Endline Household Survey will be completed among a random sample of women selected from all of the facilities' catchment areas (N= approximately 8,000). This survey will ask questions about basic demographic information, reproductive health information, HIV status, distance to the nearest health facility, prior VFP use, VFP use during project implementation, prior cervical cancer screening and preventive therapy (CCSPT) services received, and any CCSPT services received during project implementation.

ELIGIBILITY:
Inclusion Criteria:

Health care providers In-Depth Interviews (IDIs) and Focus Group Discussions:

* Health care staff member must be currently working at one of the 16 health facilities selected for the study.

Client In-Depth Interviews:

* Woman must have participated in cervical cancer screening via HPV self-sampling through one of the 16 health facilities during the study period.

Client Exit Surveys:

* Woman who received or declined VFP and/or CCS services in the catchment area of the targeted facilities.

Endline Household survey:

* Woman must be between the ages of 15-50 years.

Exclusion Criteria:

Endline Household survey:

* Woman who has had her cervix removed.

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Woman must be between the ages of 15-50 years
Enrollment: 8174 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2021-12-18 (Actual)

PRIMARY OUTCOMES:
Proportion of women who receive cervical cancer screening in Model 2 | 12 months after model implementation
  Effectiveness of community-based cervical cancer screening as measured through Endline Household Surveys
Proportion of women who receive family planning services in Model 2 | 12 months after model implementation
  Effectiveness of integrating community-based cervical cancer screening into family planning services as measured through Endline Household Surveys

SECONDARY OUTCOMES:
Proportion of healthcare workers who report satisfaction with providing cervical cancer services | 12 months after model implementation
  Acceptability and feasibility of service provision as measured through routine assessments
Proportion of healthcare workers who report satisfaction with providing family planning services | 12 months after model implementation
  Acceptability and feasibility of service provision as measured through routine assessments
Proportion of clients who report satisfaction with cervical cancer services received at study facilities | 12 months after model implementation
  Acceptability and feasibility of cervical cancer screening and preventive therapy as measured through client exit surveys
Proportion of clients who report satisfaction with family planning services received at study facilities | 12 months after model implementation
  Acceptability of family planning services as measured through client exit surveys
Cost of the intervention | 12 months after model implementation
  The cost per client of adding cervical cancer screening and preventive therapy to voluntary family planning services in each model as measured through routine assessments and client exit surveys

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tang, MD, MSCR, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Project-Malawi, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: Yes
Research data that documents, supports, and validates research findings will be made available after the main findings from the final research dataset have been accepted for publication. Access to databases will be available for educational, research, and non-profit purposes. All data to be shared will be stripped of any potentially identifying information. Data will be made available through USAID's Data Development Library (DDL).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 6 months of publication for an unlimited period
Access Criteria: Deidentified data will be publicly available through the DDL. Research datasets may also be made available to Malawian and other international investigators who request access. Requests will be evaluated on a case-by-case basis by the study investigators.
  Investigators proposing to use the data will be asked to provide approval from an ethical review committee and may be asked to execute a data use/sharing agreement with UNC. Data may be shared electronically via password protected files.
  All data sharing will abide by rules and/or policies defined by USAID, relevant IRBs, U.S. local, state, and federal laws and regulations, as well as Malawian laws and regulations. Data sharing mechanisms will ensure that the rights and privacy of individuals participating in research will be protected at all times.

REFERENCES:
- [Derived] Tang JH, Smith JS, McGue S, Gadama L, Mwapasa V, Chipeta E, Chinkhumba J, Schouten E, Ngwira B, Barnabas R, Matoga M, Chagomerana M, Chinula L. Prevention of cervical cancer through two HPV-based screen-and-treat implementation models in Malawi: protocol for a cluster randomized feasibility trial. Pilot Feasibility Stud. 2021 Apr 20;7(1):98. doi: 10.1186/s40814-021-00839-7. PMID 33879259

DOCUMENTS (1):
  • Informed Consent Form (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT04286243/ICF_000.pdf